CLINICAL TRIAL: NCT04119531
Title: Insomnia and Wake up and Recovery From Anesthesia
Status: Completed | Type: Observational
Sponsor: Adana City Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Tuna Şahin, Specialist of Anesthesiology and Reanimation, Adana City Training and Research Hospital
Record Dates: First submitted 2019-10-03; First posted 2019-10-08 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Insomnia
Keywords: anesthesia; recovery; insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with insomnia: In the preoperative room patients will be asked to participate to the study and will be asked to answer the 4-item Jenkins-Sleep Questionaire.If they accept to participate, written informed consent will be taken from the patients. According to their answers to the questionaire , patients will be divided into two groups :those with or without insomnia.
- Patients without insomnia: In the preoperative room patients will be asked to participate to the study and will be asked to answer the 4-item Jenkins-Sleep Questionaire.If they accept to participate, written informed consent will be taken from the patients. According to their answers to the questionaire , patients will be divided into two groups :those with or without insomnia.

SUMMARY:
18-55 years old 100 patients, who are planned to undergo for planned ureteroscopy will be participated in the study. In the preoperative room patients will be asked to participate to the study. If they accept 4 item Jenkins-Sleep Questionaire will be asked to them.Patients will be divided to two groups , with or without insomnia according to their answers to the questionaire. General anesthesia will be performed to all patients. At the end of operation anesthesia time,operation time, time of eye opening, time of transfer to the recovery room will be recorded in the operating room. Pain scores and recovery scores will be evaluated in the recovery room.

DETAILED DESCRIPTION:
18-55 years old 100 patients with American Society of Anesthesiology (ASA) physical status I-II,who are planned to undergo for elective ureteroscopy will be participated in this study.In the preoperative room patients will be asked to participate to the study and will be asked to answer the 4-item Jenkins-Sleep Questionaire.If they accept to participate, written informed consent will be taken from the patients. According to their answers to the questionaire , patients will be divided into two groups :those with or without insomnia.General anesthesia will be performed to all patients. After anesthesia induction with propofol 2mg/kg and rocuronium 0.6 mg/kg, patients will be ıntubated and mechanically ventilated. Maintenance of anesthesia will be achieved with 4-6 % desflurane in nitrous oxide/ oxygen (50%/50%) concentrations with the flow 5L/min. Tramadol 1 mg/kg and metoclopramid 1 ampul will be administered intravenously after intubation. Hemodynamic parameters( systolic blood pressure, diastolic blood pressure, heart rate and peripheral oxygen saturation), end tidal carbon dioxide values, the concentrations of inspired and exhaled desflurane will be recorded on the surgery start time and on the 5th, 15th,25th,35th,45th,60 th minutes of surgery. At the end of operation ,neuromuscular blockage will be reversed with neostigmine (0,05 mg/kg)and atropine sulphate 0,015 mg/kg i.v. Anesthesia time, surgery time, time of eye opening,time of transfer to the recovery room will be recorded in the operating room. In the recovery room pain score will be evaluated with Visual Analogue Scale. Modified Aldrete Recovery Score will be used for evaluating recovery.

ELIGIBILITY:
Inclusion Criteria:

* 18- 55 years
* ASA 1-2 patients
* Patients undergoing elective ureteroscopy

Exclusion Criteria:

* Renal failure
* Obstructive Sleep Apnea Syndrome,
* Thyroid dysfunction
* Neurologic and physiatric dysfunctions,
* Morbid obesity
* Anticonvulsant, antidepressant, anxiolytic drugs usage

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 18-55 years old 100 patients with American Society of Anesthesiology (ASA) physical status I-II,who are planned to undergo for elective ureteroscopy will be participated in this study.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Time of eye opening | up to 15 minutes
  from the time anesthesia was discontinued and neuromuscular blockage was reversed to the time of eye opening
Time of transpher to the postoperative care unit | up to 25 minutes
  from the time anesthesia was discontinued and neuromuscular blockage was reversed to the time of transpher to the postoperative care unit
Recovery scores | during 1 hour at postoperative period
  Modified Aldrete Recovery Score

SECONDARY OUTCOMES:
Pain scores | during 1 hour at postoperative period
  Visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Tuna Şahin, Principal Investigator — Adana City Training and Research Hospital
Locations (1):
- Tuna Şahin, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No